CLINICAL TRIAL: NCT03253926
Title: Effect of Lorcaserin on Cannabis Withdrawal and Self-administration
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Margaret Haney, Professor of Neurobiology (in Psychiatry) at CUMC, New York State Psychiatric Institute
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 7475
Record Dates: First submitted 2017-08-14; First posted 2017-08-18 (Actual); Results first posted 2022-07-26 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Cannabis Use
MeSH Terms: interventions — lorcaserin; nabiximols

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lorcaserin + Marijuana (Experimental)
  Interventions: Drug: Lorcaserin; Drug: Marijuana
- Placebo + Marijuana (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: Marijuana

INTERVENTIONS:
Drug: Lorcaserin — Lorcaserin 10mg BID
  Arms: Lorcaserin + Marijuana
Drug: Placebo — Placebo capsule BID
  Arms: Placebo + Marijuana
Drug: Marijuana — Smoked marijuana cigarette

SUMMARY:
In this study, the investigators are interested in testing how lorcaserin influences the effects of cannabis in a human laboratory model of cannabis use.

DETAILED DESCRIPTION:
In order to improve treatment outcome for cannabis use disorder (CUD), the investigators have developed a laboratory model to investigate the effects of potential treatment medications on cannabis withdrawal and on the subjective and reinforcing effects of cannabis in non treatment-seeking cannabis smokers. In this study, the investigators are interested in testing how lorcaserin influences the effects of cannabis in a human laboratory model of cannabis use.

ELIGIBILITY:
Inclusion Criteria:

* Current cannabis use
* Able to give informed consent and perform study procedures
* Women practicing an effective form of birth control
* English speaking

Exclusion Criteria:

* Presence of any clinically significant medical diagnoses
* History of heart disease and cardiac risk factors, severe chronic obstructive pulmonary disease, uncontrolled hypertension, or diabetes
* Current parole or probation
* Certain psychiatric diagnoses
* Current pregnancy or lactation

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in this study comprising two 13-day inpatient phases, each of which was preceded by two medication administration outpatient days to achieve steady-state levels prior to key behavioral measures. Each phase tested a different medication condition (lorcaserin 10 mg or placebo BID) in a within-subject design, with at least one medication-free week between phases to allow for medication clearance.
Groups:
- Lorcaserin + Marijuana First, Then Placebo + Marijuana; Placebo + Marijuana First, Then Lorcaserin + Marijuana: Lorcaserin: Lorcaserin 10mg or 0mg BID
  Marijuana: Smoked marijuana cigarette
Period: Overall Study
Arm/Group | Lorcaserin + Marijuana First, Then Placebo + Marijuana | Placebo + Marijuana First, Then Lorcaserin + Marijuana
Started | 7 | 8
Completed | 7 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Lorcaserin + Marijuana: Lorcaserin: Lorcaserin 10mg or 0mg BID
  Marijuana: Smoked marijuana cigarette
Arm/Group | Lorcaserin + Marijuana
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.9 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 2
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Cannabis Self-administration
Description: Number of cannabis puffs participant chooses to smoke.
Time Frame: 14 days
Population: Participants were randomly counterbalanced into each condition, such that all participants contributed to all conditions.
Measure: Mean (Standard Error); unit: puffs of cannabis chosen
Arm/Group | Lorcaserin + Marijuana | Placebo + Marijuana
Number analyzed (Participants) | 15 | 15
puffs of cannabis chosen
  Cannabis relapse: choice of cannabis puffs following 3 days of abstinence | 5.75 (1) | 9.2 (1)
  Cannabis abstinence initiation: choice of cannabis puffs following 0 days of abstinence | 5.75 (1) | 7.5 (1)

ADVERSE EVENTS:
Time Frame: Data reflect the number of participants reporting an adverse event during the inpatient phase (11 days) as a function of lorcaserin dose (0 mg or 10 mg BID). No serious adverse events were reported.
Arm/Group | Lorcaserin + Marijuana | Placebo + Marijuana
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 15/15 | 8/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lorcaserin + Marijuana (N=15) | Placebo + Marijuana (N=15)
Headache (Product Issues) | 3 (5) | 1 (1)
Gastrointestinal upset (Product Issues) | 6 (11) | 4 (4)
Body pain (Product Issues) | 1 (1) | 1 (1)
Anxiety/Jittery (Product Issues) | 1 (1) | 1 (1)
Eye dryness/discomfort (Product Issues) | 2 (4) | 1 (1)
Trouble sleeping (Product Issues) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
There are several limitations to consider in the current study. First, given the study length, only one dose of lorcaserin was tested, though it was the FDA-approved therapeutic dose for obesity and the dose shown to reduce tobacco cigarette use in a clinical study targeting this population. Second, the sample comprised mostly men, limiting the generalizability of our conclusions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2018-06-12): https://cdn.clinicaltrials.gov/large-docs/26/NCT03253926/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-29): https://cdn.clinicaltrials.gov/large-docs/26/NCT03253926/SAP_004.pdf
  • Informed Consent Form (2017-08-09): https://cdn.clinicaltrials.gov/large-docs/26/NCT03253926/ICF_002.pdf